CLINICAL TRIAL: NCT04129775
Title: A Randomized, Double-blind, Placebo-controlled Phase 1/2 Study of OTO-413 Given as a Single Intratympanic Injection in Subjects With Speech-in-noise Hearing Impairment
Brief Title: OTO-413 in Subjects With Speech-in-Noise Hearing Impairment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 413-201901
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Sensorineural Hearing Loss
Keywords: hearing loss; speech-in-noise; synaptopathy; hearing impairment; hidden hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss; Hearing Loss, Hidden

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTO-413 (Experimental)
  Interventions: Drug: OTO-413
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OTO-413 — Single intratympanic injection of Brain-Derived Neurotrophic Factor (BDNF)
  Arms: OTO-413
Drug: Placebo — Single intratympanic injection of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and exploratory efficacy of OTO-413 administered as an intratympanic injection for the treatment of speech-in-noise hearing impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has audiometrically-defined normal hearing or up to moderately severe hearing impairment.
* Subject has self-reported difficulty hearing in noisy environments for at least 6 months prior to Screening.
* Subject exhibited a speech-in-noise hearing deficit in at least one ear.

Exclusion Criteria:

* Subject is pregnant or lactating.
* Subject has the following hearing disorders or any other hearing disorders that may impact the efficacy assessments or safety of the subject in the opinion of the Investigator: Meniere's disease, congenital hearing loss, or genetic sensorineural hearing loss.
* Subject has a cochlear implant or consistently uses a hearing aid.
* Subject has worked at least 5 years as a professional musician or has had at least 15 years of formal musical training.
* Subject self-reports bothersome, subjective tinnitus and is consistently aware of their tinnitus throughout much of the waking day.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (Safety) | Reported or observed during or after dosing (Day 1) up to the end of study (Day 85 - 12 weeks after dosing)
  An adverse event (AE) is any unfavorable and unintended diagnosis, symptom, sign, syndrome or disease which occurs during the study, having been absent at baseline, or if present at baseline, appears to worsen.
Otoscopic Examinations (Safety) | After dosing (Day 1) up to end of study (Day 85 - 12 weeks after dosing)
  Clinically significant change form Baseline
Audiometry (Safety) | After dosing (Day 1) up to end of study (Day 85 - 12 weeks after dosing)
  Clinically significant change from Baseline

OTHER OUTCOMES:
Speech-in-noise Hearing Tests | Screening, Baseline, 2 weeks (dependent on dose group), 4 weeks, 8 weeks and 12 weeks after dosing
  Ability to hear over noise
Electrophysiological Endpoint (dependent on dose group) | At Screening, 4 weeks, 8 weeks and 12 weeks after dosing
  Electrophysiological test of auditory brainstem response to auditory stimuli
Patient Global Impression of Change | At 2 weeks (dependent on dose group), 4 weeks, 8 weeks and 12 weeks after dosing
  Change in overall hearing status, ranging from very much worse (-3) to very much improved (+3)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Colorado Otolaryngology Associates LLC dba Colorado ENT & Allergy, Colorado Springs, Colorado
  - Research Centers of America, Hollywood, Florida
  - South Florida ENT Associates or Research Centers of America, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Advanced ENT and Allergy, PLLC, Louisville, Kentucky
  - Piedmont Ear, Nose & Throat Associates, Winston-Salem, North Carolina
  - JBR Clinical Research, Salt Lake City, Utah
  - Eastern Virginia Medical School, Department of Otolaryngology, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No